CLINICAL TRIAL: NCT01238640
Title: Bioequivalence Between Two New Oral Nicotine Replacement Therapy Products and Nicorette® Microtab. A Study in Healthy Smokers
Brief Title: Bioequivalence Between Two New Oral Nicotine Replacement Therapy Products and Nicorette® Microtab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NICTDP1072; 2008-002788-15 (EudraCT Number)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Code STD (Experimental): An experimental 2 mg nicotine product coded "STD"
  Interventions: Drug: Code STD
- Code STE (Experimental): An experimental 2 mg nicotine product coded "STE"
  Interventions: Drug: Code STE
- Nicorette Microtab (Active Comparator): A comparative 2 mg marketed nicotine product called Nicorette Microtab
  Interventions: Drug: Nicorette Microtab

INTERVENTIONS:
Drug: Code STD — 2 mg Single-dose of experimental nicotine product coded "STD"
  Other Names: Not marketed
  Arms: Code STD
Drug: Code STE — 2 mg Single-dose of experimental nicotine product coded "STE"
  Other Names: Not marketed
  Arms: Code STE
Drug: Nicorette Microtab — A comparative 2 mg Single-dose of marketed tablet
  Other Names: Nicorette® Microtab
  Arms: Nicorette Microtab

SUMMARY:
The purpose of this study is to assess the bioequivalence between two new oral nicotine replacement therapy products and Nicorette® microtab.

DETAILED DESCRIPTION:
The trial has a single-dose, randomized, crossover design and includes 84 subjects. The investigational products will be given as single doses at separate treatment visits. Periods without Nicotine Replacement Therapy (NRT), lasting for at least 36 hours, will separate treatment visits. At each treatment visit, blood for pharmacokinetic analyses will be sampled immediately before, and at 5, 10, 15, 20, 30, and 45 minutes, as well as at 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 10 hours after start of product administration. The time until complete tablet dissolution will be recorded. Subjects will also be monitored to capture any adverse events that may occur. Treatment labels will be concealed from subjects and study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 10 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overall Study
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 49
Region of Enrollment [Number; unit: participants]
  Sweden | 84

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax, which is the maximum observed plasma concentration after a dose is administered, measured in nanograms/milliliter (ng/mL)
Time Frame: During 10 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- STD 2 mg: An experimental 2 mg nicotine product coded "STD"
- STE 2 mg: An experimental 2 mg nicotine product coded "STE"
- Nicorette Microtab 2 mg: A comparative 2 mg marketed nicotine product called Nicorette Microtab
Arm/Group | STD 2 mg | STE 2 mg | Nicorette Microtab 2 mg
Number analyzed (Participants) | 81 | 82 | 82
ng/mL | 3.90 (1.35) | 4.00 (1.37) | 4.08 (1.48)

2. Primary Outcome: Area Under the Curve [AUC(0-t)]
Description: Bioavailability within the Set Period [AUC(0-t)] is the area under the plasma concentration verses time curve from start of drug administration until the time of the last measurable plasma concentration, calculated as hour * nanograms (ng) per milliliter (mL).
Time Frame: During 10 hours post-dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | STD 2 mg | STE 2 mg | Nicorette Microtab 2 mg
Number analyzed (Participants) | 80 | 82 | 82
hr*ng/mL | 12.69 (5.46) | 12.56 (5.36) | 13.01 (5.80)

3. Primary Outcome: AUC(0-∞)
Description: AUC (0-∞) is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time. It is obtained from calculating AUC (0-t) plus AUC (t-∞).
Time Frame: 10 hours post-dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | STD 2 mg | STE 2 mg | Nicorette Microtab 2 mg
Number analyzed (Participants) | 80 | 82 | 82
hr*ng/mL | 15.74 (6.33) | 15.09 (6.62) | 15.57 (7.09)

4. Secondary Outcome: Product Dissolution Time
Description: Product Dissolution Time is the time from administration until the investigational products were completely dissolved.
Time Frame: During 10 hours post-dose
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | STD 2 mg | STE 2 mg | Nicorette Microtab 2 mg
Number analyzed (Participants) | 82 | 83 | 82
Minutes | 23.3 (8.90) | 23.8 (10.22) | 25.0 (6.33)

ADVERSE EVENTS:
Arm/Group | STD 2 mg | STE 2 mg | Nicorette Microtab 2 mg
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/84
Other Adverse Events (participants affected / at risk) | 11/84 | 12/84 | 19/84
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | STD 2 mg (N=84) | STE 2 mg (N=84) | Nicorette Microtab 2 mg (N=84)
Nausea (Gastrointestinal disorders) | 4 | 3 | 9
Nasopharyngitis (Infections and infestations) | 6 | 4 | 5
Headache (Nervous system disorders) | 1 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes